CLINICAL TRIAL: NCT04443127
Title: Virtual Reality as a Motor Priming Tool for Cognitive-Motor Rehabilitation Among Sub-Acute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Jaza Rizvi, Principal Invesitgator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JRizvi
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-Based Rehabilitation (Experimental)
  Interventions: Device: Virtual Reality Training Session
- Conventional Rehabilitation (Placebo Comparator)
  Interventions: Behavioral: Motor-Relearning Program

INTERVENTIONS:
Device: Virtual Reality Training Session — VR based motor priming intervention will be given for 16 sessions, comprising of 45 minutes, 4 times/week for the duration of 4 weeks on two VR environments.
  Arms: Game-Based Rehabilitation
Behavioral: Motor-Relearning Program — Motor-Relearning Program intervention will be given for 16 sessions, comprising of 45 minutes, 4 times/week for the duration of 4 weeks on two VR environments.
  Arms: Conventional Rehabilitation

SUMMARY:
Stroke is the second leading global cause of mortality counting for 6.5 million deaths per annum. The global prevalence of stroke is increasing with an estimated prevalence of 33 million per year, affecting 1 out of 6 individuals during their lifetime. The international data suggests the overall economic burden in Asia is projected to be increased to 1.3 Billion by 2050. Therefore, the appropriate and timely stroke intervention is required to save healthcare costs and reduce the burden of the disease. Studies have reported the effectiveness of VR intervention not only in cognitive abilities but it has found to be simultaneously effective in improving other domains as attention and coordination with motor retraining. VR combined with a newly developed concept of motor priming has shown encouraging results in improving motor control and task execution in stroke patients. Further studies are needed to analyze the impact of motor priming with VR in stroke patients on varied neurological domains; hence the present study aims to investigate the impact of VR based motor priming on sensorimotor, functional and cognitive outcomes among sub-acute stroke patients rehabilitation.

DETAILED DESCRIPTION:
A total 62 patients will be recruited in the study. After voluntary consent, all the patients will be randomly divided into Group-A and B through the envelope method of simple random sampling. Patients in Group-A will be receiving VR based motor priming intervention while Group-B patients will be receiving Motor-Relearning Program as conventional therapy. Whereas, both the groups will be given 16 sessions of their respective protocol, comprising of 45 minutes, 4 times/week for the duration of 4 weeks. Pre and post assessment will be performed for each patient on all three quantitative outcome measures i.e. FMA-UE, CAHAI-13, and MoCA. A trial will be terminated, if the patient reported fatigue of >8 out of 10 on the Visual Analogue Scale, unable to execute movements, reports pain, eye strain, or signs of volitional fatigue in hemiplegic or non-hemiplegic extremities.

ELIGIBILITY:
Inclusion Criteria:

* Male and female stroke patients aged 25-65 years
* Patients who had an ischemic or hemorrhagic stroke in sub-acute phase of < 3 months
* Mild cognitive impairment i.e. < 26 (19.0-25.2) on MoCA
* Minimum Scoring of 28 in the Motricity Index

Exclusion Criteria:

* Diagnosed visual-perceptual ailments which may restrict task execution
* Communication disorders such as aphasia or dysarthria which may impede cognitive assessment
* Comorbidities such as elevated blood pressure (>160mmhg/105 mmHg), heart diseases or chronic medical conditions
* Major or active psychological illness and pre-existing dementia

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Sensorimotor function of hemiplegic upper extremity (Pre-Treatment) | Baseline
  Sensorimotor function will be assessed through Fugl-Meyer Assessment Test where high values indicates increase in sensoimotor function
Sensorimotor function of hemiplegic upper extremity (Post-Treatment) | After 4 weeks
  Sensorimotor function will be assessed through Fugl-Meyer Assessment Test where high values indicates increase in sensoimotor function
Functional ability of hemiplegic upper extremity (Pre-Treatment) | Baseline
  Functional ability will be assessed through Chedoke Arm and Hand Activity Inventory-13 where high values indicates increase in Functional ability
Functional ability of hemiplegic upper extremity (Post-Treatment) | After 4 weeks
  Functional ability will be assessed through Chedoke Arm and Hand Activity Inventory-13 where high values indicates increase in Functional ability
Cognitive Function (Pre-Treatment) | Baseline
  Cognitive Function will be assessed using Montreal Cognitive Assessment where high values indicates increase in Cognitive Function
Cognitive Function (Post-Treatment) | After 4 weeks
  Cognitive Function will be assessed using Montreal Cognitive Assessment where high values indicates increase in Cognitive Function

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No